CLINICAL TRIAL: NCT01500811
Title: Evaluation the Side Effects of Autologous Chondrocyte Intra-articular Implantation in Patients With Severe Hip Osteoarthritis
Brief Title: Autologous Chondrocyte Intra-articular Implantation in Patients With Severe Hip Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Bone-009
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2011-01

CONDITIONS: Hip Osteoarthritis
Keywords: chondrocyte hip osteoarthritis intra articular injection
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Carboxylesterase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chondrocyte (Experimental): Patients with sever hip osteoarthritis who underwent intra articular cell injection.
  Interventions: Biological: cell injection

INTERVENTIONS:
Biological: cell injection — Intra articular injection of chondrocyte
  Other Names: chondrocyte transplantation

SUMMARY:
Hip osteoarthritis is degeneration of hip cartilage and inflammation of subchondral bone and soft tissue linings. Patients have pain, stiffness, swelling, and difficulty walking. There are treatments available to help manage these symptoms like weight loss, and analgesics. Surgery is the appropriate treatment in patients who have failed these conservative treatments. The aim of this clinical study is to assess safety of autologous cultured chondrocyte intra-articular injection and obtain its clinical results in patients with severe hip osteoarthritis.

DETAILED DESCRIPTION:
In this phase I clinical study 6 patients with severe hip osteoarthritis will be recruited. All patients will have a cartilage biopsy taken from the knee cartilage non-weight bearing zone. Chodrocytes will be extracted and cultured for 4 weeks. Patients then will receive chondrocyte injection under the guide of fluoroscopy. Patients will be evaluated post injection for 6 months at time intervals. Parameters considered being evaluated are, adverse effects, pain intensity and joint physical function and cartilage repair. These effects are measured by Visual Analogue Scale, WOMAC, Harris Hip Score questionnaire and MRI.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis diagnosed by MRI

Exclusion Criteria:

* Pregnancy or lactating
* Positive tests for HIV, HCV, HBV
* Active neurologic disorder
* End organ damage
* Uncontrolled endocrine disorder.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
joint swelling | 2 months
  Evaluation the swelling of hip joint after cell injection by physical examination.
deterioration of joint function | 2 months
  evaluation the deterioration of joint function by physical examination 2 months after injection in compare with base line(before injection)
dispenea | 1 week
  Evaluation the respiratory allergic reactions like dispenea by physical examination after cell injection.
skin rash | 1 week
  Evaluation the skin allergic reactions like skin rash by physical examination after cell injection.

SECONDARY OUTCOMES:
Quantitative changes in pain intensity | 2 months
  Evaluation the quantitative changes in pain measured by Visual Analogue Scale 2months after cell injection in compare with base line (before cell transplantation)
physical function improvement | 2 months
  Evaluation the physical function improvement Measured by WOMAC osteoarthritis index and Harris Hip Score 2 months after cell injection in compare with base line(before cell transplantation)
subchondral bone edema | 2 months
  Evaluation the subchondral bone edema by MRI after cell transplantation.
cartilage thickness | 2 months
  Evaluation the cartilage thickness by MRI after cell injection in compare with baseline (before cell injection)

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Royan Cell therapy Center; Mohsen Emadeddin, MD, Principal Investigator — scientist
Locations (1):
- Royan Institute, Tehran, Iran